CLINICAL TRIAL: NCT02789904
Title: Evaluation of High Sensitivity Troponin I (hsTnI) in the Management of Patients With Chest Pain in the Emergency Department
Brief Title: Evaluation of hsTnI in the Management of Patients With Chest Pain in the Emergency Department
Acronym: hsTnI
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore General Hospital (Other); Beckman Coulter GmbH (Industry); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014/2182
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2018-10

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chest pain patients in DEM: Recruitment done at SGH DEM. Blood taking will be done at 0, 1 and 2 hr.
  Interventions: Other: blood taking

INTERVENTIONS:
Other: blood taking — Blood taking will be done for chest pain patients presenting with chest pain at 0, 1 and 2 hour

SUMMARY:
Current standard of care algorithm using high sensitivity troponin T (hsTnT) requires up to 6.5 hours to diagnose an ACS. Data will be stratified based upon time of symptom onset and gender. A health economics and outcome model will be applied using the optimal high sensitivity troponin I (hsTnI) cut-off values and draw times to determine the cost and outcome benefits predicted from optimal utilization of hsTnI.

A chest pain registry will be set up to compare high sensitivity troponin I (hsTnI) versus high sensitivity troponin T (hsTnT) for all patients who present to the emergency department and require a blood draw. The outcomes of these patients will be tracked over the study period.

The purpose of conducting this study evaluation is:

1. To shorten the chest pain protocol for suitable patients to < 3 hours compared to the current 6 hours protocol with the latest high sensitivity Troponin I assays.
2. To determine the validity of Abbott ARCHITECT i2000 and Beckman Coulter ACCESS AccuTnI+3 with an accelerated algorithm in comparison to the standard of care acute coronary syndrome (ACS) algorithm and high sensitivity troponin T (hsTnT) assay, to rule-out or rule-in for an ACS within 3 hours of presentation to the emergency room (ER) with isolated suspected ACS.
3. To establish the local reference norms for hsTnI assays.

DETAILED DESCRIPTION:
Purpose

Current standard of care algorithm using high sensitivity troponin T (hsTnT) requires up to 6.5 hours to diagnose an ACS. Data will be stratified based upon time of symptom onset and gender. A health economics and outcome model will be applied using the optimal high sensitivity troponin I (hsTnI) cut-off values and draw times to determine the cost and outcome benefits predicted from optimal utilization of hsTnI.

A chest pain registry will be set up to compare high sensitivity troponin I (hsTnI) versus high sensitivity troponin T (hsTnT) for all patients who present to the emergency department and require a blood draw. The outcomes of these patients will be tracked over the study period.

The purpose of conducting this study evaluation is:

1. To shorten the chest pain protocol for suitable patients to < 3 hours compared to the current 6 hours protocol with the latest high sensitivity Troponin I assays.
2. To determine the validity of Abbott ARCHITECT i2000 and Beckman Coulter ACCESS AccuTnI+3 with an accelerated algorithm in comparison to the standard of care acute coronary syndrome (ACS) algorithm and high sensitivity troponin T (hsTnT) assay, to rule-out or rule-in for an ACS within 3 hours of presentation to the emergency room (ER) with isolated suspected ACS.
3. To establish the local reference norms for hsTnI assays.

Additionally, this study will also seek to validate the use of a 3-D Vector ECG system developed by Ngee Ann Polytechnic, to see whether improved sensitivity and specificity for the diagnosis of myocardial infarction on ECG can be achieved using vectorcardiography rather than conventional 12-lead ECG recordings.

2.0 Scope

Under the current clinical algorithm at Singapore General Hospital, ambulatory chest pain patients (CPP) receive an initial evaluation upon presentation to the ER that includes an ECG and blood draw. The lab spins and holds the blood to await add-on orders for cardiac markers if clinically-indicated. Other chest pain patients arriving by ambulance may have ECG taken in the ambulance and the results faxed ahead to the ER. Those that have an initial ECG consistent with an ST-elevation myocardial infarction (STEMI) receive immediate intervention. Patients that do not have STEMI identified are evaluated by an ER physician as soon as possible for clinical signs and symptoms of ACS, as well as, other diagnoses that require clinical treatment and/or hospital admission. Patients with suspected ACS require serial Troponin measurements as essential information for the rule-in or rule-out of a non-ST elevation myocardial infarction (NSTEMI). After seeing the patient, the ER physicians will add-on an hsTnT measurement to the sample drawn at presentation and held in the lab. This second hsTnT value is drawn two hours after presentation. Using the current standard of care hsTnT assay and the universal definition, an acute MI at Singapore General Hospital is defined as a troponin rise and/or fall with at least one value above 30pg/mL with symptoms suggestive of myocardial ischemia. There is no clear definition of the amount of rise or fall that is required. The reference range for a single troponin T measurement at Singapore General Hospital is currently defined as abnormal if above 30pg/mL. This study will compare the ARCHITECT hsTnI assay and Beckman Coulter ACCESS AccuTnI+3 assays using respective Abbott ARCHITECT and Beckman Coulter UniCel DxI 800 immunoassay systems, with hsTnT using Roche analyzer.

Troponin I is a sensitive marker of myocardial necrosis, which will be elevated due to an intraluminal coronary thrombus related to atherosclerotic plaque rupture or other spontaneous coronary artery disease (CAD) event (MI Type I). STEMI patients will be excluded from this study. The scope of this study will be limited to the rule-in and rule-out of NSTEMI in ER patients with suspected ACS and no other known causes for elevated troponin.

Healthcare data sets and Singapore General Hospital cost data will be used to assess the cost impact of an alternative model for NSTEMI diagnosis with a more aggressive hsTnI algorithm. A 30 day, Year 1, 2 and 5 follow-up phone contact in conjunction with medical record review and screening data will be used by cardiologists to determine diagnosis and confirm patient outcome.

Non-ST Elevation Myocardial Infarctions (NSTEMIs) have subtle changes in morphologies that may not be obvious on a 12-lead ECG. This limits the 12-lead ECG's ability to affirmatively indicate the presence or absence of NSTEMIs. The 3-D Vector ECG system developed by Ngee Ann Polytechnic, which has similarities to vector cardiography (VCG, i.e. the Frank lead system) is postulated to have better sensitivity to MI than the routine 12-lead ECG. Modern graphical user interface techniques used by the 3-D Vector ECG system makes interpretation easier than VCG. Additionally, since the electrode placements are identical to a 12-lead ECG. The clinical procedure for acquiring the signals is not disrupted, increasing its viability for integration into existing workflow.

3.0 Study Design and Procedures

Chest pain patients will be identified and consented in the ER waiting area following initial triage and exclusion of STEMI and within 1 hour of initial blood draw at presentation. For chest pain registry, coordinators will also invite NHCS inpatients to participate. The Clinical Coordinators, under the guidance of Study Team investigators, will be responsible to identify appropriate study candidates to join this study. They will assist the study team investigators to explain the purpose of the study and obtain informed consent for additional blood draws as well as a follow-up telephone/ medical records outcome survey. Patients will be invited to join a registry where details regarding their clinical findings, relevant investigations and clinical outcomes will be stored for possible future reference in a database. Additionally, patients will also be asked if a 6-minute ECG can be performed on them. The Clinical Coordinators will perform the 3 phlebotomy draws, which must occur within the following window periods after the presentation draw to be included in the study:

Draw Window period after presentation draw 0h 0-30 min

1. h 60-90 min
2. h 120 - 150 min

Specimens will be collected in 5.0 ml Gel tubes (Serum Separator Tube). A total of approximately 15 ml of blood will be collected from each patient. The blood sample will be processed at National Heart Centre Singapore (NHCS) laboratory. The clinical coordinators will store each patient's serum into 2 separate vials and freeze them in the freezer at ≤-80°C. The frozen serum samples will be used to perform the hsTnI assays on the Abbott ARCHITECT i2000 analyzer in NHCS and the ACCESS AccuTnI+3 assays on the Beckman Coulter UniCel Dxl 800 analyzer in SGH Pathology by the study coordinator and SGH Pathology lab staff respectively.

The screening Case Report Form is required for completion and will gather information on 3 key elements: 1) chest pain onset/characteristics; 2) comprehensive demographics to describe the study population; and 3) data for TIMI risk score generation (Appendix I).

To assess the use of 3D-Vector ECG, a target of 1000 12-lead ECGs are to be retrieved from the electrocardiographs at SGH Emergency Department triage, with the post-analysis to be done at NHCS. The retrieved ECGs will be converted to 3D-vector ECG and analysed to extract discriminating parameters which can be reliably used to diagnose and localise the presence of ischaemia. Accuracy of the diagnoses will be counter checked with the results of further diagnostic tests performed on the patient in the normal course of treatment. From the analysis of these 1000 records, the sensitivity and specificity of the 3D-Vector ECG to localise acute coronary syndrome will be computed.

4.0 Lab Test Orders, Blood Draws, and Analysis

After clinical assessment of the patient by an ER physician, an add-on troponin may be ordered for clinical purposes by the physician that will be applied to the time zero "presentation" blood draw. Likewise, a 2-hour troponin may be ordered for clinical purposes.

Analysis of Beckman Coulter ACCESS AccuTnI+3 assays will take place on UniCel DxI 800 immunoassay system in the Singapore General Hospital (SGH) Pathology. Analysis of ARCHITECT hsTnI assay will take place on Abbott ARCHITECT i2000 analyzer in the National Heart Centre Singapore (NHCS) Laboratory. Calibration, Calibration verification, cross-over validation, and daily Quality Control for the hsTnI assay will be performed by medical technologists in conjunction with normal laboratory operations.

6.0 Study Duration

4,000 patients are expected to have been included in the study in a period of 5 years from the day of recruitment. Recruitment of new patients will end after 4,000 patients are enrolled.

7.0 Data Retrieval

Laboratory data will be stored in the SingHealth Information System. Extraction of the data will be accomplished by export to an Excel spreadsheet. Clinical data will be printed out and entered into a computer database using a standardized case report form.

8.0 Telephone/ Medical records Follow-up

Study patients will be contacted by telephone/ medical records on Day 30, Year 1, Year 2 and Year 5 after recruitment for any clinical events or symptoms that will be relevant to adjudication.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 years and above
2. Ability to provide written, informed consent
3. Presentation to ER with chief complaint of chest pain OR has symptoms suggestive of angina equivalent without chest pain
4. ER physician determines patient has symptoms suggestive of ACS
5. ER physician orders troponin test for clinical purposes

Exclusion Criteria:

1. Diagnosed with STEMI
2. Poor pre-morbid Eg. Bedridden
3. Advanced malignancy/ terminal disease

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with chest pain to SGH DEM
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
First cardiovascular event | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tan Wei Chieh Jack, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No